CLINICAL TRIAL: NCT02419547
Title: Inducibility and Stability of Ventricular Tachycardia in Patients With Structural Heart Disease Undergoing VT Ablation Under General Anesthesia (Pilot Study)
Brief Title: Inducibility and Stability of Ventricular Tachycardia Inpatients Undergoing VT Ablation Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Douglas Shook, Chief, Divison of Cardiac Anesthesia, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2013-P-000241
Record Dates: First submitted 2014-09-10; First posted 2015-04-17 (Estimated); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Ventricular Tachycardia
Keywords: Ventricular tachycardia; ventricular tachycardia ablation; effects of anesthesia on VT induction; programed stimulation
MeSH Terms: conditions — Tachycardia, Ventricular | interventions — Midazolam; Fentanyl; Propofol; Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anesthesia Induction (Other): Patients undergoing ventricular tachycardia ablation will undergo programmed stimulation (PS) with minimal sedation (Versed, Fentanyl), with intravenous agents (propofol) , and finally with volatile inhalational agent (sevoflurane).
  Interventions: Drug: Versed; Drug: Fentanyl; Drug: Propofol; Drug: Sevoflurane

INTERVENTIONS:
Drug: Versed — Phase 1: Standard induction of controled sedation with intravenous agent then programed stimulation to induce ventricular tachycardia
  Other Names: midazolam
Drug: Fentanyl — Phase 1: Standard induction of controled sedation with intravenous agent then programed stimulation to induce ventricular tachycardia
  Other Names: Duragesic
Drug: Propofol — Phase 2: Standard induction of GETA with intravenous agent then programed stimulation to induce ventricular tachycardia
  Other Names: Diprivan
Drug: Sevoflurane — Phase 3: Standard induction of GETA with inhalent agent then programed stimulation to induce ventricular tachycardia
  Other Names: Ultane

SUMMARY:
This research study is being done to see whether general anesthesia (GA) affects our ability to start ventricular tachycardia (VT) during an VT ablation procedure.

Data collected during this research study will help electrophysiologists and anesthesiologists to make the best decisions about the best anesthetic conditions to use to perform VT ablations.

This research study is a "pilot" study. Pilot studies are done on a small group of subjects to learn if a larger study would be useful.

ELIGIBILITY:
Inclusion Criteria:

* Patients with VT and have an implanted ICD who are scheduled for VT catheter ablation.
* Patients 18 years of age or older

Exclusion Criteria:

* Patients with difficult airway management or patients with contra/ relative contra indication for general anesthesia or known allergies to any of the proposed anesthetic agents
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2014-07; Primary Completion 2015-04-26 (Actual); Study Completion 2015-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy L Gross, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigahm and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects undergoing VT ablation were enrolled over 1 year period
Period: Overall Study
Arm/Group | Anesthesia Induction
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Anesthesia Induction
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Had Inducible Ventricular Tachycardia Under General Anesthesia.
Description: Patients before induction of GA undergo noninvasive programmed stimulation (NIPS) using the patient's ICD. Subjects receive minimal versed/fentanyl during the NIPS. The anesthesiologist will decide whether to use propofol prior to the second induction, depending on the patient's cardiac function and hemodynamic status. After induction of GA with IV propofol, programmed stimulation will be performed from the RV catheter. Mapping under volatile agent will commence any time after twice the redistribution half-life of either agent has elapsed (propofol 4-16 mins) or have passed. Once the drug is out of the central compartment it is unlikely to affect myocardial electrolytes or ion channels. GA will be maintained with an inhalation agent, sevoflurane. A repeat programmed stimulation test will be performed. Endpoint for programmed stimulation will be induction of sustained monomorphic VT (SMVT).
Time Frame: While under General Anesthesia, an average of 6 hours
Population: All participants who underwent general anesthesia and programed stimulation during VT ablation.
Measure: Number; unit: participants
Groups:
- Ventriuclar Tachycardia Induction: Patients undergoing ventricular tachycardia ablation will undergo programmed stimulation (PS) with minimal sedation (Versed, Fentanyl), with intravenous agents (propofol) , and finally with volatile inhalational agent (sevoflurane).
  Versed: Phase 1: Standard induction of controled sedation with intravenous agent then programed stimulation to induce ventricular tachycardia
  Fentanyl: Phase 1: Standard induction of controled sedation with intravenous agent then programed stimulation to induce ventricular tachycardia
  Propofol: Phase 2: Standard induction of GETA with intravenous agent then programed stimulation to induce ventricular tachycardia
  Sevoflurane: Phase 3: Standard induction of GETA with inhalent agent then programed stimulation to induce ventricular tachycardia
Arm/Group | Ventriuclar Tachycardia Induction
Number analyzed (Participants) | 11
participants
  Phase 1 Concious Sedation | 7
  Phase 2 Propofol | 5
  Phase 3 Sevoflurane | 5

ADVERSE EVENTS:
Time Frame: 30 days
Description: There will be a 7 day follow up phone call and a 30 day visit to assess for AE's.
Arm/Group | Anesthesia Induction
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anesthesia Induction (N=11)
hematoma not requiring blood transfusion (Surgical and medical procedures) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No